CLINICAL TRIAL: NCT06576687
Title: Understanding the Neurophysiology of Ankle Instability to Improve Rehabilitation Outcomes
Brief Title: Neurophysiology of Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0549-24-EP
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-05

CONDITIONS: Ankle Injuries
Keywords: neurocognitive; neurophysiology; chronic ankle instability
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled into one of three groups based on ankle instability: mechanical instability, functional ankle instability and Coper (sprained ankle, but no residual symptoms as a comparison). Participants will complete a 4-week balance training protocol. Prior to and following the training protocol the following tasks will be completed to evaluate the training: patient-reported functioning in daily life and sports, neurocognitive hop-testing, force-control, and functional near-infrared spectroscopy (fNIRS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Balance Training (Experimental): Exercises include (1) single-limb hops to stabilization, (2) hop to stabilization and reach, (3) unanticipated hop to stabilization, (4) single-limb stance activities, and (5) continuous choice-reaction hopping.
  Interventions: Other: Physical Rehabilitation

INTERVENTIONS:
Other: Physical Rehabilitation — Exercises include (1) single-limb hops to stabilization, (2) hop to stabilization and reach, (3) unanticipated hop to stabilization, (4) single-limb stance activities, and (5) continuous choice-reaction hopping.
  Other Names: Balance and hop-training

SUMMARY:
Chronic ankle instability (CAI) is a common debilitating orthopedic condition that disrupts physical function and decreases quality of life. Not all CAI is the same. It can be mechanical ligamentous laxity, perceived disability often referred to as functional instability, or a combination of the two. However, clinicians and researchers most often combine all chronic ankle instability patients without considering these sub-groups, which may account for poor recovery and recurrence. The objective of this research is to determine functional and neurophysiological differences between sub-groups of CAI to allow for development of evidence-based rehabilitation which may improve patient outcomes.

To accomplish this, the study will determine the differences among CAI sub-groups on performance of a traditional side-hop test and neurocognitive hop test, determine differences in neurophysiological response and motor control between CAI sub-groups during a lower limb and an ankle specific task, and determine the underlying neurophysiological effects of a 4-week neurocognitively enhanced balance training protocol among CAI subgroups. Time to complete each of the hop tests, cortical activation during the balance and force control tasks, and neurocognitive performance will be assessed to determine differences in performance and neurological function among subgroups of CAI

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is a common debilitating orthopedic condition that disrupts physical function and decreases quality of life. CAI is heterogenous and can manifest as mechanical ligamentous laxity, perceived disability often referred to as functional instability, or a combination of the two. However, clinicians and researchers most often combine all chronic ankle instability patients without considering these sub-groups, which may account for the poor recovery and recurrent nature of this pathology. Neurocognitive and neurophysiologic discrepancies may explain the different sub-groups; however, technological limitations have previously limited this assessment. The objective of this research is to determine functional and neurophysiological differences between sub-groups of CAI to allow for development of evidence-based rehabilitation which may improve patient outcomes.

To accomplish this, the study will determine the differences among CAI sub-groups on performance of a traditional side-hop test and neurocognitive hop test, determine differences in neurophysiological response and motor control between CAI sub-groups during a lower limb and an ankle specific task, and determine the underlying neurophysiological effects of a 4-week neurocognitively enhanced balance training protocol among CAI subgroups. This study hypothesizes functional performance will be similar between sub-groups during a traditional side-hop test, but those with functional instability without mechanical laxity will perform worse during a choice-reaction hop test compared to those with mechanical ankle instability. It also hypothesizes individuals with functional ankle instability will demonstrate greater cortical activation during the research tasks and after a 4-week balance training protocol compared to individuals with mechanical ankle instability. Time to complete each of the hop tests, cortical activation during the balance and force control tasks, and neurocognitive performance will be assessed to determine differences in performance and neurological function among subgroups of CAI.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be physically active (participation in at least 90 total minutes of activity/week including running, walking, lifting weights, or playing a sport, etc.)
* Healthy controls:

  * no history of lateral ankle sprain
  * no complaints of their ankle giving way
  * a Cumberland Ankle Instability Tool (CAIT) score greater than 28
* Coper participants (participants coping with ankle problems:

  * a history of lateral ankle sprain, but no episodes of giving way in previous 12 months
  * CAIT score greater than 28
* Chronic ankle instability (CAI):

  * history of ankle sprain
  * two or more episodes of ankle giving way in previous 12 months
  * CAIT score less than 25

Exclusion Criteria:

* History of lower extremity surgery or fracture
* Current signs or symptoms of a joint sprain in the lower extremity
* Pregnancy
* Diagnosis of a vestibular disorder
* Diagnosis of a nerve or connective tissue disorder
* Significant history of condition that impaired cognitive function such as concussion or learning disability
* Currently taking medications that may affect cognitive function such as narcotics, anti-depressants, anti-anxiety agents, or stimulants

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Side-hop Test | Baseline and post-rehabilitation (six weeks total)
  Amount of time it takes participants to hop medially and laterally across a 30-cm gap ten times will be measured. Greater times equals worse performance.
Choice-reaction Hop Test | Baseline and post-rehabilitation (six weeks total)
  Amount of time it takes participants hop on a mat medially and laterally across a 30-cm gap ten times, using visual cues to direct movement to one of two squares on each side. Greater times equals worse performance.
Inversion-eversion Force Control | Baseline and post-rehabilitation (six weeks total)
  The force control accuracy at 50% maximal contraction for eversion and inversion will be determined. This is analyzed by a non-linear analysis Lyapunov exponent (LyE) which measures the quality or the natural, inherent fluctuations in movement. Greater values indicate reduced neuromuscular control.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool | Baseline and post-rehabilitation (six weeks total)
  Cumberland Ankle Instability Tool (CAIT), a 9-item scale, will be used to measure the severity of functional ankle instability. It is scored from 0 to 30. Higher scores indicate a better outcome.
Foot and Ankle Ability Measure Activities of Daily Living (FAAM-ADL) Scale | Baseline and post-rehabilitation (six weeks total)
  The Foot and Ankle Ability Measure Activities of Daily Living Scale will be used to assess physical function in activities of daily living (ADL) for individuals with foot and ankle impairments. It is a patient-reported outcome instrument that is scored as a percentage from 0% to 100%. Higher scores indicate a better outcome.
Foot and Ankle Ability Measure Sport (FAAM-Sport) Scale | Baseline and post-rehabilitation (six weeks total)
  The Foot and Ankle Ability Measure Activities of Daily Living Scale will be used to assess physical function in sports activities for individuals with foot and ankle impairments. It is a patient-reported outcome instrument that is scored as a percentage from 0% to 100%. Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adam B Rosen, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska-Omaha, Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No